CLINICAL TRIAL: NCT02970136
Title: Increasing Uptake of Evidence-Based Screening Services Through CHW-led Multi-modality Intervention: South Florida Center for Reducing Health Disparities
Brief Title: Increasing Uptake of Evidence-Based Screening Services Through CHW-led Multi-modality Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Olveen Carrasquillo, Professor of Medicine and Public Health Sciences, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: 20160023; 1U01MD010614-01 (NIH)
Record Dates: First submitted 2016-11-18; First posted 2016-11-21 (Estimated); Results first posted 2021-12-28 (Actual); Last update posted 2021-12-28 (Actual); Status verified 2021-11

CONDITIONS: Human Papillomavirus; Human Immunodeficiency Virus; Hepatitis C; ColoRectal Cancer
Keywords: Increased Screening Uptake; Community Health Worker; Medically Underserved
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome; Hepatitis C; Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Home Based Screening (Experimental): The participant will be receiving home-based screening tests (OraQuick Swab, OraQuick Fingerstick, Human Papillomavirus (HPV) Self-Sampling Test, Fecal Immunochemical Test) delivered by the community health worker
  Interventions: Device: OraQuick Swab; Device: Fecal Immunochemical Test; Device: OraQuick Fingerstick; Device: HPV Self-Sampling Test; Other: Home Based Screening Tests
- Clinic Based Screening (Active Comparator): The participant will meet the Community Health Worker and will be navigated to a clinic appointment for standard screening tests
  Interventions: Other: Standard Screening Tests

INTERVENTIONS:
Device: OraQuick Swab — OraQuick for oral fluid HIV antibody testing
  Arms: Home Based Screening
Device: Fecal Immunochemical Test — Fecal Immunochemical stool test specific for human hemoglobin
  Arms: Home Based Screening
Device: OraQuick Fingerstick — Patients will be tested for Hepatitis C infection using a fingerstick
  Arms: Home Based Screening
Other: Standard Screening Tests — Patients will be navigated to a local health center for standard screening tests
  Arms: Clinic Based Screening
Device: HPV Self-Sampling Test — Patients will be using swab to check for HPV infection
  Arms: Home Based Screening
Other: Home Based Screening Tests — Patients will provided screening tests and instructed by Community Health Worker on how to perform home screening tests
  Arms: Home Based Screening

SUMMARY:
The purpose of this research study is to determine the best way to increase screening for cervical cancer, colorectal cancer, HIV, and Hepatitis C among under screened Hispanic, Haitian and African-American individuals in Hialeah, South Dade, and Little Haiti. The investigator will compare home testing led by a community health worker (CHW) versus clinic testing guided by a CHW. Community Health Workers are people who have undergone several weeks of community outreach and health education training. During the study period the participant will continue to receive all of their regular medical care from their regular health care providers. If the participant does not have a health care provider, the Community Health Workers would be able to help in referring the participant for care at a local health care clinic located in their community.

ELIGIBILITY:
Inclusion Criteria:

1. live in one of the three target communities
2. self-identify as Haitian, Hispanic and/or Black.
3. be 50-64 years old
4. need at least one of the four recommended screening services as per US Preventive Service Task Force 121 guidelines as follows: never having had a HIV test b) never having had a Hepatitis C Virus (HCV) test c) not having a Pap smear in the last three years d) not having had a colonoscopy in last 10 years and/or stool-based test in the last year.

Exclusion Criteria:

1. plan to move out of the community during the next six months;
2. current or prior enrollment (5 five years) in any research study that involved screening for these conditions.
3. Are adults unable to consent
4. Are individuals who are not yet adults (infants, children, teenagers)
5. Pregnant women
6. Prisoners

Ages: 50 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 754 (Actual)
Dates: Start 2017-04-11 (Actual); Primary Completion 2020-10-30 (Actual); Study Completion 2020-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Olveen Carrasquillo, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Carrasquillo O, Seay J, Jhaveri V, Long T, Kenya S, Thomas E, Sussman D, Trevil D, Koru-Sengul T, Kobetz E. Increasing uptake of evidence-based screening services though a community health worker-delivered multimodality program: study protocol for a randomized pragmatic trial. Trials. 2020 Apr 29;21(1):368. doi: 10.1186/s13063-020-4213-7. PMID 32349789

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Home Based Screening | Clinic Based Screening
Started | 377 | 377
Completed | 297 | 282
Not Completed | 80 | 95

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Home Based Screening | Clinic Based Screening | Total
Number analyzed (Participants) | 377 | 377 | 754
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.33 (4.54) | 57.40 (4.49) | 57.37 (4.51)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 282 | 282 | 564
  Male | 95 | 95 | 190
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 239 | 241 | 480
  Not Hispanic or Latino | 138 | 136 | 274
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 142 | 143 | 285
  White | 205 | 214 | 419
  More than one race | 28 | 19 | 47
  Unknown or Not Reported | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Are Screened for All Conditions
Description: As evaluated by participant self report and completed sampling kits. Female participants are to be screened on 4 conditions: HIV, HCV, Human Papilloma Virus (HPV) and Fecal Immunochemical Testing (FIT). Male participants are to be screened on 3 conditions: HIV, Hepatitis C Virus (HCV) and FIT.
Time Frame: Baseline
Population: There were 282 female participants and 95 male participants enrolled for each arm for a total of 377 total enrolled participants per arm. Female participants are to be screened on 4 conditions: HIV, HCV, Human Papilloma Virus (HPV) and Fecal Immunochemical Testing (FIT). Male participants are to be screened on 3 conditions: HIV, Hepatitis C Virus (HCV) and FIT.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Home Based Screening | Clinic Based Screening
Number analyzed (Participants) | 377 | 377
Percentage of participants
  Female Participants: number analyzed (Participants) | 282 | 282
  Female Participants | 25.18 [20.22 to 30.24] | 8.16 [5.24 to 11.99]
  Male Participants: number analyzed (Participants) | 95 | 95
  Male Participants | 32.63 [23.36 to 43.02] | 15.79 [9.02 to 24.70]

2. Secondary Outcome: Change in Percentage of Participants Completing Screening Test From Baseline to 6 Months
Description: As evaluated by participant self report and completed sampling kits. Female participants are to be screened on 4 conditions: HIV, HCV, HPV and FIT. Male participants are to be screened on 3 conditions: HIV, HCV and FIT.
Time Frame: Baseline, Up to 6 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Home Based Screening | Clinic Based Screening
Number analyzed (Participants) | 377 | 377
percentage of participants
  HCV Screening Test | 71.88 [67.35 to 76.42] | 31.56 [26.87 to 36.26]
  HIV Screening Test | 46.15 [41.12 to 51.19] | 20.95 [16.85 to 25.06]
  HPV Screening Test: number analyzed (Participants) | 282 | 282
  HPV Screening Test | 24.47 [19.45 to 29.49] | 12.06 [8.26 to 15.86]
  FIT Screening Test | 39.26 [34.33 to 44.19] | 18.57 [14.64 to 22.49]

3. Secondary Outcome: Median Number of Screenings Completed
Description: as for outcome 2
Time Frame: At baseline and at 6 months
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: screenings completed
Arm/Group | Home Based Screening | Clinic Based Screening
Number analyzed (Participants) | 377 | 377
screenings completed
  Female Participants at Baseline: number analyzed (Participants) | 282 | 282
  Female Participants at Baseline | 1 [1 to 2] | 1 [0 to 2]
  Female Participants at 6 months: number analyzed (Participants) | 282 | 282
  Female Participants at 6 months | 4 [2 to 4] | 2 [1 to 3]
  Male participants at Baseline: number analyzed (Participants) | 95 | 95
  Male participants at Baseline | 1 [0 to 1] | 1 [0 to 1]
  Male Participants at 6 months: number analyzed (Participants) | 95 | 95
  Male Participants at 6 months | 3 [2 to 3] | 2 [1 to 3]

ADVERSE EVENTS:
Time Frame: Up to 6 months
Arm/Group | Home Based Screening | Clinic Based Screening
All-Cause Mortality (participants affected / at risk) | 0/377 | 0/377
Serious Adverse Events (participants affected / at risk) | 0/377 | 0/377
Other Adverse Events (participants affected / at risk) | 0/377 | 0/377

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-11): https://cdn.clinicaltrials.gov/large-docs/36/NCT02970136/Prot_SAP_000.pdf